CLINICAL TRIAL: NCT01829360
Title: Interactive Book Reading to Accelerate Word Learning by Children With SLI
Brief Title: Accelerating Word Learning in Children With Language Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01DC012824 (NIH); R01DC012824 (NIH)
Record Dates: First submitted 2013-03-12; First posted 2013-04-11 (Estimated); Results first posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-10

CONDITIONS: Specific Language Impairment
MeSH Terms: conditions — Specific Language Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants that collect and score the pre/post outcomes are blind to arm assignment.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard then Alternative: High Dose (Experimental): Children in this arm are assigned to the standard treatment for the first round of intervention (dose 6 x dose frequency 6) and then the alternative treatment that maximizes dose (dose 9 x dose frequency 4)
  Interventions: Behavioral: Treatment (interactive book reading, dialogic reading, shared book reading)
- Alternative: High Dose then Standard (Experimental): Children in this arm are assigned to the alternative treatment that maximizes dose (dose 9 x dose frequency 4) in the first round of intervention and then to the standard treatment for the second round of intervention (dose 6 x dose frequency 6)
  Interventions: Behavioral: Treatment (interactive book reading, dialogic reading, shared book reading)
- Alternative: High Dose Frequency then Standard (Experimental): Children in this arm are assigned to the alternative treatment that maximizes dose frequency (dose 4 x dose frequency 9) in the first round of intervention and then to the standard treatment for the second round of intervention (dose 6 x dose frequency 6)
  Interventions: Behavioral: Treatment (interactive book reading, dialogic reading, shared book reading)
- Standard then Alternative: High Dose Frequency (Experimental): Children in this arm are assigned to the standard treatment for the first round of intervention (dose 6 x dose frequency 6) and then the alternative treatment that maximizes dose frequency (dose 4 x dose frequency 9)
  Interventions: Behavioral: Treatment (interactive book reading, dialogic reading, shared book reading)

INTERVENTIONS:
Behavioral: Treatment (interactive book reading, dialogic reading, shared book reading) — Children receive 2 rounds of treatment with interactive book reading. Each treatment teaches 30 words that the children do not know. Treatments vary in dose (the number of times the words is heard/taught in an individual book reading session: 4 vs. 6 vs. 9) and dose frequency (the number of times book reading sessions are repeated: 4 vs. 6. vs. 9). Across all dose x dose frequency combinations, children hear/are taught the 30 words 36 times, which has been shown to be the adequate overall intensity of the intervention.
  Other Names: Interactive book reading; Dialogic reading; Shared book reading

SUMMARY:
This research attempts to adapt and optimize a word learning treatment, specifically interactive book reading, for use with Kindergarten children with Specific Language Impairment (SLI). Children with SLI have difficulty learning language without any obvious cause for this difficulty. This study will examine the best way to achieve the appropriate intensity of 36 exposures. For example, is it better to hear the new words many times within the book (high dose) and to read the book few times (low dose frequency), or is it better to hear the new words a few times within the book (low dose) and to read the book many times (high dose frequency). The investigators hypothesize that reading the books many times will be more effective than repeating the words many times within a book.

DETAILED DESCRIPTION:
Specific Language Impairment (SLI) affects approximately 7.4% of Kindergarten children. Children with SLI are known to have difficulty learning new words, which places them at greater risk for future reading impairments and academic failure. Surprisingly, there are few interventions for word learning by children with SLI that have undergone rigorous efficacy and/or effectiveness testing. The goal of this research is to optimize an interactive book reading intervention that has proven to be successful in teaching vocabulary to other groups of Kindergarten children. A secondary goal was to examine whether pre-treatment characteristics predicted how many words children would learn.

This study further tests the adequate intensity of 36 exposures. Each child will receive two treatments at the identified adequate intensity. Children were randomized to two treatments: the standard treatment and 1 of 2 alternative treatments. The standard treatment used in prior research was balanced between the amount of times the new word is heard within the book (dose 6) and the amount of times the book is read (dose frequency 6). The alternative treatments were more heavily weighted for either repetitions within the book (high dose/low dose frequency, i.e., dose 9 x dose frequency 4) or the amount of times the book is read (low dose/high dose frequency, i.e., dose 4 x dose frequency 9). Ultimately, this study determines how best to achieve the adequate intensity of 36 exposures.

A secondary goal was to further examine the pre-treatment factors associated with the number of words learned by children with SLI during interactive book reading. We once again explore a variety of potential predictors including those that were significant in a prior study (i.e., phonological awareness, nonword repetition, and semantics) as well as those that were not significant in a prior study but that had the potential to be related to a child's ability to learn during interactive book reading. That is, a child's general language abilities (as measured by the Clinical Evaluation of Language Fundamentals-4, CELF-4, Core Language score) and their ability to understand verbally presented stories (as measured by the CELF-4 Understanding Spoken Paragraphs score) could impact their success in encoding new words during interactive book reading.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Kindergarten enrollment
* Age 5 to 6 years
* Normal hearing
* Nonverbal Intelligence Quotient (IQ) of 85 or higher on the Reynolds Intellectual Assessment Scale
* Score below 82 on the Clinical Evaluation of Language Fundamentals
* Score at or below the 10% percentile on one of the approved standardized vocabulary assessments.

Exclusion Criteria:

* Speaks more than one language
* Health history indicating neurologic or other disorder that would exclude a diagnosis of SLI (e.g., autism, developmental disability, seizure disorder)

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Storkel, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Treatment & Testing Scripts — http://doi.org/10.23641/asha.9745181 — See item S4 and S7.

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Then Alternative: High Dose: Treatment 1= dose 6 x dose frequency 6 Treatment 2 = dose 9 x dose frequency 4
- Alternative: High Dose Then Standard: Treatment 1= dose 9 x dose frequency 4 Treatment 2 = dose 6 x dose frequency 6
- Alternative: High Dose Frequency Then Standard: Treatment 1= dose 4 x dose frequency 9 Treatment 2 = dose 6 x dose frequency 6
- Standard Then Alternative: High Dose Frequency: Treatment 1= dose 6 x dose frequency 6 Treatment 2 = dose 4 x dose frequency 9
Period: Overall Study
Arm/Group | Standard Then Alternative: High Dose | Alternative: High Dose Then Standard | Alternative: High Dose Frequency Then Standard | Standard Then Alternative: High Dose Frequency
Started | 8 | 9 | 10 | 8
Completed | 8 | 9 | 9 | 8
Not Completed | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Alternative: High Dose Frequency Then Standard: Treatment 1= dose 4 x dose frequency 49 Treatment 2 = dose 6 x dose frequency 6
- Total: Total of all reporting groups
Arm/Group | Standard Then Alternative: High Dose | Alternative: High Dose Then Standard | Alternative: High Dose Frequency Then Standard | Standard Then Alternative: High Dose Frequency | Total
Number analyzed (Participants) | 8 | 9 | 9 | 8 | 34
Age, Continuous [Mean (Standard Deviation); unit: months] | 65 (3) | 68 (4) | 68 (4) | 64 (4) | 66 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 1 | 13
  Male | 4 | 5 | 5 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 7 | 9 | 8 | 30
  Unknown or Not Reported | 2 | 1 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 3
  White | 6 | 7 | 8 | 8 | 29
  More than one race | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 9 | 8 | 34
Target Vocabulary Probe [Mean (Standard Deviation); unit: Number correct] — The average number of correctly defined words for each of the two word sets that will be taught during the two rounds of treatment. Number of words correct can range from 0 to all 30 words in a set. On average, children new approximately 0-1 word prior to treatment (range 0-5 words).
  Number correct
    Treatment 1: Pre | 0.63 (0.92) | 0.78 (0.67) | 0.56 (0.88) | 0.38 (0.52) | 0.59 (0.74)
    Treatment 2: Pre | 0.63 (0.74) | 0.56 (0.73) | 1.44 (1.59) | 0.38 (0.52) | 0.76 (1.05)

OUTCOME MEASURES:

1. Primary Outcome: Change in Words Known From Pre- to Post-treatment
Description: In each of the two treatments, children are taught 30 new words and tested on their ability to provide a definition of each word. Definitions are scored as 0 points for an incorrect or absent definition, 1 point for an appropriate use of the word in a sentence or for a vague definition, 2 points for a conventional definition containing at least one critical element but lacking other critical elements, and 3 points for a complete and accurate definition including all critical elements. For the analyses, children's definitions scored as 2 or 3 (i.e., a partially or completely accurate definition) were counted as correct (i.e., the child knows the word) and definitions scored as 0 or 1 (i.e., incorrect definition, absent definition, correct use of a word in a sentence, or vague definition) were counted as incorrect (i.e., the child does not know the word). Thus, children's scores could range from 0 to 30 words known, with higher scores indicating better outcomes.
Time Frame: Pre- and Post-treatment with treatment lasting 10 to 23 sessions (approximately 5 to 12 weeks)
Measure: Mean (Standard Error); unit: Number of words learned
Groups:
- Standard Then Alternative: High Dose: Treatment 1 = dose 6 x dose frequency 6 Treatment 2 = dose 9 x dose frequency 4
- Alternative: High Dose Then Standard: Treatment 1 = dose 9 x dose frequency 4 Treatment 2 = dose 6 x dose frequency 6
- High Dose Frequency Then Standard: Treatment 1 = dose 4 x dose frequency 9 Treatment 2 = dose 6 x dose frequency 6
- Standard Then Alternative: High Dose Frequency: Treatment 1 = dose 6 x dose frequency 6 Treatment 2 = dose 4 x dose frequency 9
Arm/Group | Standard Then Alternative: High Dose | Alternative: High Dose Then Standard | High Dose Frequency Then Standard | Standard Then Alternative: High Dose Frequency
Number analyzed (Participants) | 8 | 9 | 9 | 8
Number of words learned
  Treatment 1: Pre | 0.63 (0.32) | 0.78 (0.22) | 0.56 (0.29) | 0.38 (0.25)
  Treatment 1: Post | 6.88 (1.82) | 2.44 (0.77) | 3.67 (1.39) | 2.75 (0.70)
  Treatment 2: Pre | 0.63 (0.26) | 0.56 (0.24) | 1.44 (0.53) | 0.38 (0.18)
  Treatment 2: Post | 4.13 (0.52) | 3.67 (1.05) | 5.89 (2.14) | 4.75 (1.22)
Statistical Analysis 1: Comparison: Standard Then Alternative: High Dose vs Alternative: High Dose Then Standard vs High Dose Frequency Then Standard vs Standard Then Alternative: High Dose Frequency; Test type: Superiority; p < 0.05, Mixed Models Analysis; The significance of fixed effects (e.g.,treatment) was evaluated using Wald tests
Statistical Analysis 2: Comparison: Standard Then Alternative: High Dose vs Alternative: High Dose Then Standard vs High Dose Frequency Then Standard vs Standard Then Alternative: High Dose Frequency; Test type: Other — A secondary analysis was performed to examine individual differences in treatment outcomes. This was done collapsed across all arms because the difference between the arms/treatments was not significant in the primary analysis. This was done by adding predictors to the primary analysis model to determine if learner characteristics were significantly related to growth in word defining. All continuous learner characteristics were grand mean centered; p < 0.05, Mixed Models Analysis

2. Secondary Outcome: Interim Definition
Description: Learning also was tracked during treatment. The research assistant who provided the treatment prompted children to provide definitions at four points during each treatment. Depending on the arm, the four test points corresponded to 6-9 exposures, 18-20 exposures, 27-30 exposures, and 36 exposures.The words were assessed in a fixed order while the child viewed the pre-reading pictures for each word. The research assistant asked, "What does [word] mean?". Specific feedback was not provided but the correct definition always was provided after the child's response regardless of the accuracy of the response. Scoring was the same as that described for definitions administered pre/post. Scores could range from 0-30 words correctly defined.
Time Frame: Treatment lasted 5-12 weeks. Data was taken during this time.
Measure: Mean (Standard Error); unit: Number of words correct
Arm/Group | Standard Then Alternative: High Dose | Alternative: High Dose Then Standard | Alternative: High Dose Frequency Then Standard | Standard Then Alternative: High Dose Frequency
Number analyzed (Participants) | 8 | 9 | 9 | 8
Number of words correct
  Treatment 1: Test 1 | 3.00 (0.73) | 5.11 (1.05) | 6.33 (1.52) | 5.38 (0.65)
  Treatment 1: Test 2 | 12.13 (1.44) | 8.00 (1.55) | 9.67 (2.04) | 8.13 (1.66)
  Treatment 1: Test 3 | 9.25 (2.10) | 9.89 (1.49) | 10.33 (2.26) | 10.13 (1.87)
  Treatment 1: Test 4 | 10.13 (1.57) | 10.00 (1.42) | 12.78 (2.49) | 10.13 (2.32)
  Treatment 2: Test 1 | 4.25 (0.88) | 6.44 (0.82) | 4.56 (1.03) | 4.75 (1.16)
  Treatment 2: Test 2 | 6.00 (1.43) | 9.00 (1.55) | 8.22 (1.75) | 6.25 (1.59)
  Treatment 2: Test 3 | 9.13 (1.46) | 11.22 (1.37) | 9.00 (2.04) | 6.38 (1.82)
  Treatment 2: Test 4 | 9.00 (2.04) | 9.78 (1.91) | 10.67 (1.99) | 9.50 (1.88)
Statistical Analysis 1: Comparison: Standard Then Alternative: High Dose vs Alternative: High Dose Then Standard vs Alternative: High Dose Frequency Then Standard vs Standard Then Alternative: High Dose Frequency; The interim definition data were analyzed with the primary pre-/post-definition data to capture growth across the entire treatment period; Test type: Superiority; p < 0.05, Mixed Models Analysis

3. Secondary Outcome: Interim Naming
Description: Learning also was tracked during treatment. The research assistant who provided the treatment prompted children to name the target words at four points during each treatment. Depending on the arm, the four test points corresponded to 6-9 exposures, 18-20 exposures, 27-30 exposures, and 36 exposures. The research assistant showed the child the post-book reading picture without the orthographic label and asked a question meant to elicit the phonological form of the target word (e.g., "What is the lightning doing?" to elicit flashing). Specific feedback was not provided but the correct orthographic label and context sentence always were provided after the child's response regardless of the accuracy of the response. Responses were scored as correct (i.e., matched the target word) or incorrect (i.e., did not match the target word). Total score could range from 0 to 30 words correctly named in each treatment.
Time Frame: Administered during treatment, which lasted 5-12 weeks
Measure: Mean (Standard Error); unit: Number of words correct
Arm/Group | Standard Then Alternative: High Dose | Alternative: High Dose Then Standard | Alternative: High Dose Frequency Then Standard | Standard Then Alternative: High Dose Frequency
Number analyzed (Participants) | 8 | 9 | 9 | 8
Number of words correct
  Treatment 1: Test 1 | 0.63 (0.26) | 0.78 (0.46) | 0.44 (0.18) | 0.38 (0.26)
  Treatment 1: Test 2 | 3.88 (1.51) | 1.44 (1.00) | 4.67 (1.33) | 2.88 (1.06)
  Treatment 1: Test 3 | 5.63 (1.89) | 2.89 (1.35) | 6.44 (1.66) | 6.00 (1.50)
  Treatment 1: Test 4 | 5.50 (2.12) | 3.67 (1.51) | 6.56 (1.74) | 8.00 (2.32)
  Treatment 2: Test 1 | 0.38 (0.38) | 0.67 (0.24) | 0.44 (0.24) | 1.50 (0.42)
  Treatment 2: Test 2 | 2.25 (0.70) | 2.67 (1.12) | 3.00 (1.38) | 5.75 (1.82)
  Treatment 2: Test 3 | 4.50 (1.78) | 4.67 (1.52) | 5.67 (1.99) | 7.75 (2.23)
  Treatment 2: Test 4 | 7.38 (2.65) | 7.33 (2.40) | 7.44 (2.59) | 10.88 (1.80)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during study participation. Children engaged in two rounds of treatment with each round lasting 5-12 weeks, depending on arm assignment. In addition, post-treatment data was collected approximately 1-week after treatment ended. Thus, the entire monitoring period was 11-25 weeks for each participant, depending on arm.
Description: Definition does not differ.
Arm/Group | Standard Then Alternative: High Dose | Alternative: High Dose Then Standard | High Dose Frequency Then Standard | Standard Then Alternative: High Dose Frequency
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
No limitations noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT01829360/Prot_SAP_000.pdf